CLINICAL TRIAL: NCT02820155
Title: A Double-Blind, Randomized, Placebo-Controlled, Dose-Escalating, Single Dose and Multiple Dose Study to Evaluate the Safety and Pharmacokinetics of RGN1016 in Healthy Male Subjects
Brief Title: Phase I Single and Multiple Escalating Dose Study of RGN1016 in Healthy Male Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201412002MIPD
Record Dates: First submitted 2016-06-03; First posted 2016-06-30 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
Keywords: Alzheimer's disease,cognitive function
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo (Placebo Comparator): Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Interventions: Drug: Placebo
- RGN1016_50mg (Experimental): Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Interventions: Drug: RGN1016
- RGN1016_100mg (Experimental): Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Interventions: Drug: RGN1016
- RGN1016_200mg (Experimental): Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Interventions: Drug: RGN1016
- RGN1016_400mg (Experimental): Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Interventions: Drug: RGN1016
- RGN1016_800mg (Experimental): Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Interventions: Drug: RGN1016

INTERVENTIONS:
Drug: RGN1016 — Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Arms: RGN1016_100mg; RGN1016_200mg; RGN1016_400mg; RGN1016_50mg; RGN1016_800mg
Drug: Placebo — Stage I: single oral dose Stage II: multiple oral dose (QD, 7days)
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, dose-escalating, single dose and multiple dose study.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, dose-escalating study. The study comprises single dose (Stage I) and multiple dose (Stage II) stages. Stage II will not be initiated until completion of Stage I. The interim safety analysis report will be submitted to TFDA for an approval for proceeding to Stage II.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be entered in the study only if they meet all of the following criteria:

1. Male with suitable veins for cannulation or repeated venipuncture, and must be able to swallow the study drug intact;
2. Aged between 20 and 45 years (inclusive) at the screening visit;
3. Has normal hematology results at screening visit;

   * WBC: 3.54 ~ 9.06X10^3/μL
   * RBC: 4 ~ 5.52X10^6/μL
   * hemoglobin: 13.2 ~17.2 g/dL
   * hematocrit: 40.4 ~ 51.1%
   * platelet: 148 ~ 339X10^3/μL
4. Has normal biochemistry results at screening visit;

   * alkaline phosphatase: 34 ~ 104 U/L
   * total bilirubin: 0.3 ~ 1.0 mg/dL
   * AST: 8 ~ 31 U/L
   * ALT: 0 ~ 41 U/L
   * BUN: 7 ~ 25 mg/dL
   * creatinine: 0.6 ~ 1.3 mg/dL
5. Normal coagulation results at screening visit;

   * Prothrombin time/INR: 9.8 ~ 11.5 sec/0.92 ~ 1.09
   * PTT: 25.6~32.6 sec
6. Normal blood pressure (systolic blood pressure: 100 ~ 140 mmHg; diastolic blood pressure: 60 ~ 90 mmHg) at screening visit or prior to administration of investigational product;
7. Able to provide written informed consent and willing to comply with the study protocol procedures and restrictions.

Exclusion Criteria:

Subjects must not satisfy any of the following criteria:

1. Has a body weight less than 50 kg and/or body mass index (BMI) less than 18 kg/m^2 or greater than 30 kg/m^2 at the screening visit. Body mass index is determined as total body weight/height^2 (kg/m^2);
2. Is not in good general health as judged by the Investigator based on medical history, vital signs, physical examination, ECG, laboratory tests, and urinalysis at the screening visit or prior to administration of investigational product;
3. Has a history or presence of any disease or condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs at the screening visit or prior to administration of investigational product;
4. Has a clinically significant psychiatric, renal, hepatic, cardiovascular, gastrointestinal, or neurologic disease at screening or prior to administration of investigational product;
5. Is a smoker and/or has used nicotine-containing products within the last 6 months prior to the screening visit;
6. Has a history of alcohol and/or drug abuse;
7. Participation of any clinical investigation during the last 60 days;
8. Blood donation of more than 250 mL within the past 12 weeks;
9. Excessive intake of caffeine containing drinks or food (more than 6 units of caffeine per day). One caffeine unit is contained in the following items: 1 (177.4 mL) cup of coffee, 2 (354.9 mL) cans of cola, 1 (354.9 mL) cup of tea, ½ (118.3 mL) cup of energy drink (e.g., PAOLYTA B Liq. or WHISBIH Liq.) or 3 oz of chocolate;
10. Use of drugs with enzyme inducing properties such as St. John's Wort within 4 weeks prior to dosing;
11. Has used prescription or nonprescription medication (except for occasional use of paracetamol and nasal spray) or herbal remedies or vitamins or minerals within 2 weeks or 5 half-lives of the drug, whichever is longer, prior to dosing;
12. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of study medication;
13. Male subjects who are unwilling to use barrier contraception in addition to having their partner use another method of contraception, for the duration of the study and for 3 months after dosing;
14. Has a positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus (HIV);
15. Has received a blood transfusion within the last 6 months at screening;
16. Involved in the planning or conduct of the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Number of incidence of Adverse Events. | up to14 days

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | 8 days
Time to peak drug concentration (Tmax) | 8 days
Maximum Plasma Concentration (Cmax) | 8 days
Half-life T1/2 | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jang Chiu, Principal Investigator — Neurology department of National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided